CLINICAL TRIAL: NCT00599209
Title: Health Information Technology in the Nursing Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Baycrest Centre for Geriatric Care (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Jerry Gurwitz, MD Executive Director, Meyers Primary Care Institute/University of Massachusetts Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11390; 5R01HS015430 (AHRQ)
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Patient Safety; Prescribing Practices; Laboratory Monitoring Practices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - coded unit ID (Experimental): Nursing home units provided the CDS intervention
  Interventions: Other: clinical decision support
- B - coded unit ID (No Intervention): Nursing home units not provided the CDS intervention

INTERVENTIONS:
Other: clinical decision support — CDS is provided to prescribers on intervention units upon ordering medication which offers advice on prescribing and monitoring practices
  Arms: A - coded unit ID

SUMMARY:
The magnitude and intensity of medication use among our nation's 1.6 million nursing home residents matches or exceeds that of hospitalized patients. The residents of nursing homes are among the most frail patients in the population; the challenges of using medications in this setting are great, not only because of the physiologic declines and pharmacologic changes that occur with aging, but also because of the special clinical and social circumstances that often characterize nursing home care. In our previous research, we have determined that medication errors resulting in adverse drug events occur most often at the ordering and monitoring stages of pharmaceutical care. Clinical decision-support systems are clinical consultation systems that combine individual patient information with population statistics and scientific evidence to offer real-time information to health care providers. These systems have been found to improve the quality of medication prescribing in the hospital setting. In this study, we intend to determine the extent to which a computer-based clinical decision-support system (accompanying computerized provider order-entry) can improve the quality of medication ordering and monitoring for residents in the long-term care setting through a randomized trial. We will track the costs associated with this system and the system's impact on the productivity of providers. We will also assess the culture of U.S. nursing homes and the organization of the nursing home setting with respect to readiness to incorporate computerized provider order-entry with computer-based clinical decision support. Our project addresses specific areas that are of particular interest to AHRQ with special relevance to the delivery of high-quality care to a priority population--the frail elderly patient population residing in nursing homes. The project will assess the economic implications of health information technology in the nursing home environment that will be of interest to key stakeholders, including physicians, pharmacists, nurses, payers, policymakers, the nursing home industry, and pharmaceutical vendors to long-term care institutions.

ELIGIBILITY:
Inclusion Criteria:

* prescriber at the study facility

Exclusion Criteria:

* not a prescriber at the study facility

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
extent to which a computer-based clinical decision-support system (accompanying computerized provider order-entry) can improve the quality of medication ordering and monitoring | two years

SECONDARY OUTCOMES:
costs associated with this system and the system's impact on the productivity of providers | two years

CONTACTS AND LOCATIONS:
Overall Officials: Jerry H Gurwitz, MD, Principal Investigator — Meyers Primary Care Institute
Locations (1):
- Meyers Primary Care Institute, Worcester, Massachusetts, United States

REFERENCES:
- [Background] Subramanian S, Hoover S, Gilman B, Field TS, Mutter R, Gurwitz JH. Computerized physician order entry with clinical decision support in long-term care facilities: costs and benefits to stakeholders. J Am Geriatr Soc. 2007 Sep;55(9):1451-7. doi: 10.1111/j.1532-5415.2007.01304.x. PMID 17915344
- [Derived] Field TS, Rochon P, Lee M, Gavendo L, Baril JL, Gurwitz JH. Computerized clinical decision support during medication ordering for long-term care residents with renal insufficiency. J Am Med Inform Assoc. 2009 Jul-Aug;16(4):480-5. doi: 10.1197/jamia.M2981. Epub 2009 Apr 23. PMID 19390107